CLINICAL TRIAL: NCT06987578
Title: Osteopathic Manipulative Treatment vs. Standard Therapy in the Management of Acute Neck and Low Back Pain in the Emergency Department
Brief Title: OMT vs. Standard Therapy in the Management of Acute Neck and Low Back Pain in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Regional Medical Center, New Jersey (Other)
Collaborators: American Osteopathic Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR#19-025
Record Dates: First submitted 2022-10-17; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Acute Pain
Keywords: musculoskeletal pain
MeSH Terms: conditions — Acute Pain; Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: block randomization OMT vs Standard treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OMT only (Other): THE OMT study group will receive 5 minutes of OMT treatment consisting of either or both myofascial release and muscle energy
  Interventions: Other: OMT vs. Ibruprofen
- ibuprofen or placebo (Placebo Comparator): The control group will only receive ibuprofen 400mg in a single dose
  Interventions: Other: OMT vs. Ibruprofen

INTERVENTIONS:
Other: OMT vs. Ibruprofen — OMT vs. Standard Therapy in the Management of Acute Neck and Low Back Pain in the Emergency Department

SUMMARY:
Patients 18 to 65 years old who present within 72 hours of onset pain will be considered for study enrollment. Patients with the acute musculoskeletal low back or neck pain based on ED history and structural physical exam will be included. Patients will be excluded based upon specific exclusion criteria. After providing informed consent, patients will be randomized by block randomization to receive OMT or ibuprofen 400 mg, given orally.

DETAILED DESCRIPTION:
Patients 18 to 65 years old who present withinj 72 hours of onset pain will be considered for study enrollment. Patients with acute musculoskeletal low back or neck pain based on ED history and structural physical exam will be included. Patients will be excluded based upon specific exclusion criteria. After providing informed consent, patients will be randomized by block randomization to receive OMT or ibuprofen 400 mg, given orally.

A unique patient code will be given to each patient to protect their privacy. A baseline pain score of an 11-point numeric rating scale (NRS-11) will be documented prior to the intervention. The OMT study group will receive 5 minutes of OMT treatment consisting of either or both myofascial release and muscle energy. The control group will only receive ibuprofen 400 mg in a single oral dose. At 30 and 60 minutes post intervention both groups will be asked to score their pain on the 11-point NRS scale from 0 to 10. At 60 minutes, each patient will also be asked to evaluate their perceived pain reduction on the 5-point pain reduction scale (PRS-5). A pain reduction of 50% or greater, on the NRS-11 scale, will be considered clinically significant. Additionally patients will be asked to assess whether they experienced any significant side effects, such as nausea, vomiting, epigastric pain, dizziness or worsening muscle soreness. If the patient's pain is not controlled by 60 minutes, patients will be offered rescue analgesia. The choice of analgesic will be left to the discretion of the provider, but will be recorded for analysis. Lastly, patient satisfaction and likability of treatment will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 to 65 years old who present within 72 hours of onset pain will be considered for study enrollment. Patients with acute musculoskeletal low back or neck pain based on ED history and structural physical exam will be included, provided they sign the informed consent.

Exclusion Criteria:

* Failure to sign consent Focal neurological deficit (motor or sensory), or paresthesia

  * Severe osteoporosis
  * History of peptic ulcer disease
  * Presentation requiring cardiac monitoring
  * Fracture, dislocation, or joint instability at the area of symptoms
  * Presentation after traumatic injury requiring C-collar placement prior to or subsequent to arrival
  * Cancer or malignancy of the head, neck, chest or back
  * Allergy to aspirin or nonsteroidal anti-inflammatory drugs
  * Cellulitis (skin infection) at the treatment site
  * Pregnancy or currently breastfeeding
  * History of renal impairment
  * Cervical or lumbar radiculopathy
  * Active illicit drug abuse or chronic alcohol use
  * Chronic pain syndrome
  * Daily opioid use
  * Use of aspirin daily
  * Use of antiplatelet or anticoagulant medications (clopidogrel, warfarin, dabigatran rivaroxaban, apixaban or other similar medications)
  * Glasgow Coma Scale (GCS) less than 15 or altered mental status
  * Prisoners presenting in police custody
  * Use of any non-steroidal antiplatelet medications (NSAIDS) or administration of any non-pharmacological manipulation (Physical Therapy or OMT) within six hours prior to presentation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
decrease opiod use | 10/30/2022
OMT vs. Standard Therapy in the Management of Acute Neck and Low Back Pain in the Emergency Department | 60 minutes
  50% change in pain score on the NRS-11 pain scale, from time of randomization to 60 minutes post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Loretta Hall, MBHA, Study Director — St. Joseph's University Medical Center
Locations (1):
- St. Joseph's University Medical Cener, Paterson, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
A unique code will replace a subject identifiers